CLINICAL TRIAL: NCT04142567
Title: Role of the Clinical Pharmacist in an Oncology Ambulatory Center to Prevent Drug Related Problems Before Antitumor Treatment Initiation
Brief Title: Role of the Pharmacist in Detection of Drug Interactions Before Antitumor Treatment Initiation
Acronym: CHOPIN
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A03512-53
Record Dates: First submitted 2019-09-04; First posted 2019-10-29 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Neoplasm
Keywords: Drug drug interactions; Pharmacist interventions; Cancer patients; Out patient setting
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this observational study is to evaluate the benefits of a pharmacist integration in an oncology ambulatory center, to prevent drug related problems (in particular drug drug interactions) at antitumor treatment initiation.

The hypothesis of this work is that a drug drug interaction will be observed in 30% of cancer patients and will have a major clinical impact in 1% of the cases. The primary endpoint is the prevalence of pharmacist interventions among patients who are going to receive an oral targeted therapy or cancer chemotherapy or immunotherapy

DETAILED DESCRIPTION:
The purpose of this observational study is to evaluate the benefits of a pharmacist integration in an oncology ambulatory center, to prevent drug related problems (in particular drug drug interactions) at antitumor treatment initiation.

The hypothesis of this work is that a drug drug interaction will be observed in 30% of cancer patients and will have a major clinical impact in 1% of the cases.

The primary endpoint is the prevalence of pharmacist interventions among cancer patients who are going to receive an oral targeted therapy (140 patients) or cancer chemotherapy or immunotherapy (300 patients).

Pharmacist interventions will be classified according to the SFPC (société française de pharmacie Clinique) classification.

The secondary endpoints are

* The detection of drug drug interactions with theriaque software, Micromedex software and DDI predictor tool.
* The clinical gradation by an independent expert comity of the clinical impact of avoided drug drug interaction. The expert comity will grade avoided clinical consequences in 3 levels (minor, moderate or major),
* The Economic evaluation of pharmacist intervention: Cost of the project to evaluate drug drug interaction and benefits after evaluation of avoided clinical consequences
* The Adherence evaluation of patients treated with oral cancer targeted therapy (Therefore, only patients under oral targeted therapy will be evaluated at Day0, Day15 ,Day 30 and Month 6 to determine adherence.)

ELIGIBILITY:
Inclusion Criteria:

* legal age patients
* Affiliated to social security or with another insurance system
* with a solid tumor
* who are going to receive an antitumor treatment (chemotherapy, immunotherapy or oral targeted therapy)

Exclusion Criteria:

* pregnant women
* minor patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients in outpatient setting, treated in two Paris hospitals
Sampling Method: Non-Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
Prevalence of Pharmacist intervention | up to 1 week from date of inclusion
  Percentage of patients whom antitumora treatment or usual treatment has been changed by the pharmacist intervention

SECONDARY OUTCOMES:
Detection of Drug -drug interactions | up to 1 week from date of inclusion
  Number of drug drug interactions detected
Clinical gradation of drug drug interactions | One year
  Gradation by an independent experts comity of the clinical impact of prevented drug drug interaction
Cost of the pharmacist intervention by avoided clinical consequence | One year
  Cost evaluation of pharmacist for analysis and medication review with patient by avoided interaction
Potential cost of the avoided clinical consequences | One year
  Treatment cost of avoided clinical consequences , balanced with the probability of occurrence
Adherence evaluation with oral cancer targeted therapy by therapeutic drug monitoring | day 15, 30 and 6 months after oral therapy initiation
  Patients with plasma drug concentration below the 10th percentile will be classified as nonadherent patients
Adherence evaluation with oral cancer targeted therapy by the 6 item-Girerd Scale | day 15, 30 and 6 months after oral therapy initiation
  Patients with a Girerd score greater than or equal to 3 will be classified as nonadherent patients
Adherence evaluation with oral cancer targeted therapy by pill count | 6 months after oral therapy initiation
  Pill counts will be used to calculate the percent of total prescribed dose taken to prescribed during the 90-day period

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Thomas-Schoemann, PharmD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- APHP -Cochin Hospital and Georges Pompidou European Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thomas-Schoemann A, Blanchet B, Bardin C, Noe G, Boudou-Rouquette P, Vidal M, Goldwasser F. Drug interactions with solid tumour-targeted therapies. Crit Rev Oncol Hematol. 2014 Jan;89(1):179-96. doi: 10.1016/j.critrevonc.2013.08.007. Epub 2013 Aug 28. PMID 24041628
- [Background] P. Boudou Rouquette, A. Thomas-Schoemann, A. Chahwakilian et al., Clinical benefit of a one-day multidisciplinary work-up for risk assessment in unfit cancer patients. ESMO congress, abstract 1558; Amsterdam 2013
- [Background] Bonnet C, Boudou-Rouquette P, Azoulay-Rutman E, Huillard O, Golmard JL, Carton E, Noe G, Vidal M, Orvoen G, Chah Wakilian A, Villeminey C, Blanchet B, Alexandre J, Goldwasser F, Thomas-Schoemann A. Potential drug-drug interactions with abiraterone in metastatic castration-resistant prostate cancer patients: a prevalence study in France. Cancer Chemother Pharmacol. 2017 May;79(5):1051-1055. doi: 10.1007/s00280-017-3291-z. Epub 2017 Mar 30. PMID 28361167
- [Background] Lees J, Chan A. Polypharmacy in elderly patients with cancer: clinical implications and management. Lancet Oncol. 2011 Dec;12(13):1249-57. doi: 10.1016/S1470-2045(11)70040-7. Epub 2011 Jul 6. PMID 21741307
- [Background] Riechelmann RP, Tannock IF, Wang L, Saad ED, Taback NA, Krzyzanowska MK. Potential drug interactions and duplicate prescriptions among cancer patients. J Natl Cancer Inst. 2007 Apr 18;99(8):592-600. doi: 10.1093/jnci/djk130. PMID 17440160
- [Background] Ruddy K, Mayer E, Partridge A. Patient adherence and persistence with oral anticancer treatment. CA Cancer J Clin. 2009 Jan-Feb;59(1):56-66. doi: 10.3322/caac.20004. PMID 19147869